CLINICAL TRIAL: NCT02635763
Title: A Randomized Controlled Trial of Comparing Two Methods of Nerve Block in Combination With Laryngeal Mask Anesthesia Effect for Hip Fracture on Post-operative Quality of Recovery in Elderly Patients
Brief Title: Peripheral Nerve Blocks in Elderly Patients With Hip Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Qingfu Zhang, Shanghaii Sixth People's Hospital, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NB001
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Hip Fracture
Keywords: nerve block; general anesthesia; hip fracture; recovery
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PNBs1 (Other): Femoral nerve and the lateral cutaneous nerve block combined with general anesthesia
  Interventions: Procedure: Femoral nerve and the lateral cutaneous nerve block
- PNBs2 (Other): Lumbar plexus and sacral plexus nerve block combined with general anesthesia
  Interventions: Procedure: Lumbar plexus and sacral plexus nerve block

INTERVENTIONS:
Procedure: Femoral nerve and the lateral cutaneous nerve block — Femoral nerve block was performed using 0.5% ropivacaine (15ml) under ultrasound guide;the lateral cutaneous nerve block was performed using 0.5% ropivacaine (5ml) under ultrasound guide
  Arms: PNBs1
Procedure: Lumbar plexus and sacral plexus nerve block — Lumbar plexus block was performed using 0.5% ropivacaine (25ml) under ultrasound guide; sacral plexus nerve block was performed using 0.5% ropivacaine (15ml) under ultrasound guide
  Arms: PNBs2

SUMMARY:
As the population ages, the frequency of surgery is increasing proportionally, bringing with it the challenge of managing older patients with frequent comorbid diseases and an increased risk of complications. Poor postoperative quality of recovery may result in patient and family suffering, a prolonged hospital stay, and a greater demand on health care resources.The purpose of this study was to evaluate the ultrasound guided percutaneous femoral nerve+lateral cutaneous nerve versus lumbar plexus+sacral plexus nerve block composite laryngeal mask anesthesia in elderly hip fracture surgery, the application of assessing their impact on the postoperative recovery quality.

DETAILED DESCRIPTION:
In this study, patients who were more than 65 years old with hip fracture were randomized to peripheral nerve blocks 1(PNBs1)- femoral nerve+lateral cutaneous nerve-with laryngeal mask anesthesia, or peripheral nerve blocks 2(PNBs2) - lumbar plexus and sciatic - with laryngeal mask anesthesia. Blocks were performed using ultrasound and 0.5% ropivacaine. All patients received postoperative multimodal analgesia. Postoperative recovery was assessed at 15 minutes, 40 minutes,- 1 day, 3 days, and 7 days after surgery, with the Postoperative Quality of Recovery Scale, in physiological, nociceptive, emotive, modified activities of daily living, modified cognitive, and overall patient perspective domains.

ELIGIBILITY:
Inclusion Criteria:

1. ASA grade I ~ III level;
2. The BMI <30;
3. The Mini - getting the state examination MMSE > 23;
4. The operation type:open reduction and internal fixation or bipolar head replace.

Exclusion Criteria:

1. Serious systemic diseases such as respiratory dysfunction, cardiac insufficiency, and renal insufficiency;
2. Has a history of cognitive function disorder or mental illness;
3. Has a history of cerebral infarction and leave sequela;
4. The blood coagulation dysfunction;
5. The hearing or visual impairment;
6. Unable to complete assessment;
7. Operation time more than 90 minutes;
8. The bleeding is greater than 1000 ml.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
postoperative quality of recovery | 3 days after operative

CONTACTS AND LOCATIONS:
Overall Officials: Junfeng Zhang, PhD, Study Director — Department of Anesthesiology, Shanghai Jiao Tong University Affiliated Shanghai Sixth People's Hospital
Locations (1):
- Shanghai Jiao Tong University Affiliated Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Urwin SC, Parker MJ, Griffiths R. General versus regional anaesthesia for hip fracture surgery: a meta-analysis of randomized trials. Br J Anaesth. 2000 Apr;84(4):450-5. doi: 10.1093/oxfordjournals.bja.a013468. PMID 10823094
- [Background] Abou-Setta AM, Beaupre LA, Rashiq S, Dryden DM, Hamm MP, Sadowski CA, Menon MR, Majumdar SR, Wilson DM, Karkhaneh M, Mousavi SS, Wong K, Tjosvold L, Jones CA. Comparative effectiveness of pain management interventions for hip fracture: a systematic review. Ann Intern Med. 2011 Aug 16;155(4):234-45. doi: 10.7326/0003-4819-155-4-201108160-00346. PMID 21844549
- [Background] Liu J, Yuan W, Wang X, Royse CF, Gong M, Zhao Y, Zhang H. Peripheral nerve blocks versus general anesthesia for total knee replacement in elderly patients on the postoperative quality of recovery. Clin Interv Aging. 2014 Feb 18;9:341-50. doi: 10.2147/CIA.S56116. eCollection 2014. PMID 24600214